CLINICAL TRIAL: NCT06566352
Title: Different Methods to Minimize Blood Loss During Laparoscopic Myomectomy; A Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Nashat Fatah Allah Omran, Obstetrics and Gynecology Department Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 218/12-3-2024
Record Dates: First submitted 2024-08-01; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Different Methods to Minimize Blood Loss During Laparoscopic Myomectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- laparoscopic myomectomy with temporary bilateral uterine artery occlusion (Experimental): laparoscopic myomectomy with temporary bilateral uterine artery occlusion
  Interventions: Procedure: laparoscopic myomectomy with temporary bilateral uterine artery occlusion
- Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine (Experimental): Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine
  Interventions: Procedure: Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine; Drug: injection of epinephrine 1mg diluted in 200mg of NaCl
- traditional laparoscopic myomectomy (Experimental): traditional laparoscopic myomectomy
  Interventions: Procedure: traditional laparoscopic myomectomy

INTERVENTIONS:
Procedure: Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine — intramyometrial injection of epinephrine 1mg diluted in 200mg of NaCl solution
  Arms: Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine
Procedure: traditional laparoscopic myomectomy — traditional laparoscopic myomectomy
  Arms: traditional laparoscopic myomectomy
Procedure: laparoscopic myomectomy with temporary bilateral uterine artery occlusion — Experimental: laparoscopic myomectomy with temporary bilateral uterine artery occlusion
  Arms: laparoscopic myomectomy with temporary bilateral uterine artery occlusion
Drug: injection of epinephrine 1mg diluted in 200mg of NaCl — injection of epinephrine 1mg diluted in 200mg of NaCl
  Arms: Laparoscopic myomectomy with intramyometrial injection of diluted epinephrine

SUMMARY:
Laparoscopic myomectomy with temporary bilateral uterine artery occlusion or intramyometrial injection of diluted epinephrine will be important to reduce intraoperative bleeding, time of operation and hospitalization period after laparoscopic myomectomy.

DETAILED DESCRIPTION:
Laparoscopic myomectomy with temporary bilateral uterine artery occlusion or intramyometrial injection of diluted epinephrine will be important to reduce intraoperative bleeding, time of operation, and hospitalization period after laparoscopic myomectomy.

This will be the first study to investigate the efficacy of Laparoscopic myomectomy with temporary bilateral uterine artery occlusion or intramyometrial injection of diluted epinephrine in minimizing blood loss during Laparoscopic myomectomy at our university.

Can Laparoscopic myomectomy with temporary bilateral uterine artery occlusion or intramyometrial injection of diluted epinephrine give better outcomes regarding intraoperative bleeding when compared to traditional laparoscopic myomectomy?

ELIGIBILITY:
Inclusion Criteria:

1. Women aged from 18 to 39 years.
2. Symptomatizing Women (heavy menstrual bleeding or subfertility).
3. FIGO stage (3-7) by ultrasound.
4. Only uterine corpus fibroid.
5. Up to three fibroids by ultrasound.
6. No previous hormonal treatment.

Exclusion Criteria:

1. Patients with bleeding tendency.
2. Patients who refuse to participate in the study or uncooperative patients.
3. Current pregnancy.
4. Any retroperitoneal surgery at pararectal space.
5. More than one cesarean delivery.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
blood loss | intra-operative
  estimated blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided